CLINICAL TRIAL: NCT05487157
Title: Social Workers of Elderly Care in Hungary- Investigation of Workplace Conditions- Workplace Stress, Burnout and Turnover Intention After the Covid-19 Pandemic
Brief Title: Social Workers of Elderly Care in Hungary
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: BMEÜ/599-3/2022/EKU
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2023-08

CONDITIONS: Stress; COVID-19; Burnout, Professional
Keywords: social workers; stress; turnover; covid-19; burnout; hungarian social sector; validation of TIS
MeSH Terms: conditions — COVID-19; Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Actively employed social workers in Hungary: Eligibility criteria: Social workers in Hungary, who are actively employed, 18 years of age or older, working in the field of elderly care.
  Exclusion criteria: people, who do not have an active employment; currently have no job; working online; non-professional staff working in social care (eg. cleaning, maintenance)

SUMMARY:
In our Research the goal is to examine the level of stress and burnout among social care workers and their causes and effects after COVID-19 pandemic. We would like to examine the migration from work trend and its socio-demographic causes in the light of COVID-19 pandemic among social care workers in Hungary. We would like to analyze the extent of stress and burnout at work after COVID-19 pandemic, as well as the resulting turnover intentions in Hungary among social care workers. Our goal is to validate on hungarian population the Turnover Intention Scale (TIS-6), to measure fluctuation and migration.

DETAILED DESCRIPTION:
A number of stress factors have been identified that affect nurses' burnout and job change, but there is little domestic research on the topic among social workers in connection with the COVID-19 epidemic.

As a result of our research, we expect that higher fear of COVID-19 is associated with lower job satisfaction, increased workplace anxiety, burnout, and increased turnover intentions.

ELIGIBILITY:
Inclusion Criteria:

* Social workers in Hungary, who are actively employed,
* 18 years of age or older
* working in the field of elderly care.

Exclusion Criteria:

* people, who do not have an active employment
* currently have no job
* working online
* non-professional staff working in social care (eg. cleaning, maintenance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hungarian actively employed Social workers
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Social workers's stress, burnout and turnover intention | Day 1
  Measure the level of stress, burnout and turnover intention after COVID-19 Pandemic
Social workers's stress, burnout and turnover intention | Day 1
  Validate on hungarian population the Turnover Intention Scale (TIS-6), to measure fluctuation and migration.
  The 6-question version of the TIS questionnaire evaluates the answers on a 5-point Likert Scale. The midpoint of the scale is 18 (3 x 6). If the total score is below 18 then the it indicates a desire to stay. If the scores are above 18 it indicates a desire to leave the organisation. The minimum a person can get is 6 (6 x 1) and the maximum is 30 (5 x 6). No item scores need to be reflected (reverse scored) for the TIS-6.

CONTACTS AND LOCATIONS:
Locations (1):
- Overall Hungary, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nemeth Z, Deak P, Makai A, Hock M. Exploring the mediating effect of burnout between fear of COVID-19, job-related stress and turnover intention among elderly care workers. BMC Health Serv Res. 2025 Nov 25;25(1):1526. doi: 10.1186/s12913-025-13700-x. PMID 41291748